CLINICAL TRIAL: NCT00120354
Title: Long-Term Lamivudine Therapy for Chronic Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050195; 05-DK-0195
Record Dates: First submitted 2005-07-15; First posted 2005-07-15 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-03-31

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B Virus; Antiviral Resistance; Drug Withdrawal; Immune Response; Hepatitis B Surface Antigen; Liver Biopsy; Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B; Substance Withdrawal Syndrome | interventions — Hematologic Tests

INTERVENTIONS:
Procedure: Blood Testing
Procedure: Percutaneous Liver Biopsy
Procedure: Lamivudine Therapy

SUMMARY:
This study will evaluate the long-term safety and effectiveness of lamivudine therapy and the possibility of stopping therapy in patients whose hepatitis B is chronic, that is, long lasting, and which has responded to treatment. Chronic hepatitis B, caused by a virus, is a common form of liver disease affecting about 1 million Americans and about 5 percent of the world's population. Health effects include a continuous state of being infectious and the risk of transmitting hepatitis to other people, symptoms of liver disease, and development of cirrhosis-that is, severe damage to the liver-and liver cancer. Lamivudine is a medication that blocks hepatitis B effectively but does not make it disappear completely. Scientists believe that the immune system must also be active to rid the body of the last traces of hepatitis B.

Patients ages 18 and older who have chronic hepatitis B and are being treated with lamivudine may be eligible to participate in this study. They will undergo a medical history and physical examination and will be given lamivudine in 100 mg tablets to be taken as one tablet, once each day. Patients will be asked to return to the outpatient clinic every 3 months, when they will undergo a brief interview and measurement of vital signs-such as blood pressure, pulse, and body weight. During the visits, they will fill out questionnaires about any symptoms or side effects they have, and they will be seen by a doctor and have a brief medical history and examination. There will be a collection of blood for complete blood counts, liver enzymes, and hepatitis B virus. Extra blood tests may be done to analyze patients' immune reactions to hepatitis B. Patients will also receive refills of their lamivudine tablets. They will continue to be treated with lamivudine as long as it seems to control the hepatitis infection and liver disease.

At intervals of about 1 year, patients will have ultrasound examinations, lasting about 1 hour, of the liver and abdomen. Then at intervals of about 5 years, patients will undergo liver biopsies, which require a hospital stay of 2 to 3 days. A liver biopsy is done by passing a needle through the skin into the liver to obtain a piece of liver about 2 inches long and 1/16-inch in diameter. A small amount of bleeding probably occurs with most liver biopsies. Internal bleeding is a risk, which may require that the patient stay in the hospital a few days longer, for rest, observation and pain medicine. The biopsy provides information that proves whether lamivudine is controlling the liver disease and preventing it from worsening or progressing to cirrhosis.

Side effects of lamivudine include fatigue, muscle aches, fever and chills, sore throat, nausea, stomach pain or cramps, and diarrhea. Serious side effects are rare, occurring in less than 1% of people taking lamivudine. They include inflammation of the pancreas, nerve damage, and buildup of lactic acid in the blood. About 25% of patients experience a temporary worsening, or flare, of hepatitis during the first few months of treatment. If flares are severe, it is important for researchers to determine whether they are caused by resistance to lamivudine or by the immune system acting against the hepatitis B virus or another liver condition. A flare of hepatitis can also occur when lamivudine is stopped, that is, a withdrawal. In such situations, testing for hepatitis B virus levels and other liver conditions is important. It may lead to other treatments or stopping lamivudine and taking another medication instead. While patients are participating in the study, they will have a careful evaluation of their hepatitis and general condition. They may have an improvement in their disease as a result of long-term lamivudine therapy.

DETAILED DESCRIPTION:
The major aims of this study are to evaluate the long-term efficacy and safety of lamivudine therapy and the possibility of stopping therapy in a cohort of patients with chronic hepatitis B who have a maintained response to treatment. Lamivudine is a nucleoside analogue with potent activity against hepatitis B virus (HBV), which is approved for use in the United States and is used extensively throughout the world to treat HBV and HIV infection. Lamivudine is well tolerated and adverse events are rare. Its major shortcoming is the development of antiviral resistance after prolonged therapy which results in loss of effectiveness, marked by rise in viral levels and return of disease activity. Some patients, however, have a maintained response to lamivudine therapy and in these individuals treatment is continued indefinitely or until hepatitis B surface antigen (HBsAg) is lost and therapy can be permanently stopped. This protocol will allow for the long-term treatment and evaluation of these patients. Patients will be maintained on lamivudine at a dose of 100 mg daily and seen every three months for interim medical history and serum testing for aminotransferase levels and hepatitis B markers, with liver biopsies done every 5 years. Lamivudine will be stopped if HBsAg is lost. The protocol also includes an option to attempt withdrawal of therapy under controlled conditions focusing on inducing immune reactivity to HBV and clearance of HBsAg. Patients will stop lamivudine for short periods (1 week, and later for 2, 4 and 8 weeks) and be monitored during and for 12 weeks afterwards for aminotransferase levels, HBV DNA levels and CD4+ and CD8+ T cell responses to HBV antigens. Patients who demonstrate significant worsening of hepatitis will not undergo further attempts at withdrawal. The endpoint to successful therapy is defined as loss of hepatitis B surface antigen (HBsAg) and development of antibody (anti-HBs).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18 years or above, male or female
* Presence of HBsAg in serum for at least 6 months.
* Previous liver biopsy histology showing chronic hepatitis with or without cirrhosis.
* Long-term (greater than 1 year) lamivudine therapy in doses of 100 mg daily.
* Normal or near normal (less than twice the upper limit of normal) serum aminotransferase levels.
* HBV DNA levels below 10(5) copies per ml while on lamivudine.
* Written informed consent.

EXCLUSION CRITERIA:

* In women, pregnancy, breast feeding, and, in those capable of bearing children, inability to practice adequate contraception.
* Significant systemic illnesses other than liver disease, including congestive heart failure, renal failure, chronic pancreatitis, or diabetes mellitus with poor control.
* Serum creatinine greater than 1.5 mg/dL and creatinine clearance less than 50 cc/min.
* A history of clinically apparent pancreatitis or evidence of subclinical pancreatitis as shown by serum amylase values twice the upper limits of the normal range and abnormalities of the pancreas on computerized tomography or other imaging studies of the abdomen.
* Severe cirrhosis as defined by Child's stage C (Child-Pugh score of 7 or above).
* HIV infection as indicated by presence of anti-HIV in serum.
* Chronic hepatitis C as shown by the presence of anti-HCV and HCV RNA in serum.
* Immunosuppressive therapy requiring use of more than 10 mg of prednisone (or its equivalent) per day.
* Other antiviral therapy for chronic hepatitis B within the previous 3 months.
* Sensory or motor neuropathy apparent from medical history and physical examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-07-11; Study Completion 2007-03-31

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Lok AS, McMahon BJ; Practice Guidelines Committee, American Association for the Study of Liver Diseases (AASLD). Chronic hepatitis B: update of recommendations. Hepatology. 2004 Mar;39(3):857-61. doi: 10.1002/hep.20110. No abstract available. PMID 14999707